CLINICAL TRIAL: NCT02833909
Title: ex Vivo Study of the Inflammatory Response Associated With Hidradenitis Suppurativa
Brief Title: Activation of a Cutaneous Inflammasome in the Skin of Hidradenitis Suppurativa Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PO14129
Record Dates: First submitted 2016-07-04; First posted 2016-07-14 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2016-07

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Surgical Procedures, Operative

ARMS (2):
- HS (Experimental)
  Interventions: Other: surgery
- Controls (Experimental)
  Interventions: Other: surgery

INTERVENTIONS:
Other: surgery

SUMMARY:
The objective is to investigate ex vivo the inflammatory response in hidradenitis suppurativa (HS) (activation of an inflammasome, role of pro-inflammatory cytokines) in the skin of patients treated surgically for this disease.

The investigators hypothesize that Th17-derived cytokines, especially Interleukin (IL) IL-17, could serve as a relay in the inflammatory process leading to HS severity and recurrences.

DETAILED DESCRIPTION:
The objective is to investigate ex vivo the inflammatory response in hidradenitis suppurativa (activation of an inflammasome, role of pro-inflammatory cytokines) in the skin of patients treated surgically for this disease.

The investigators hypothesize that Th17-derived cytokines, especially IL-17, could serve as a relay in the inflammatory process leading to HS severity and recurrences.To fulfil this proposal, the investigators will aim at demonstrating and characterizing the presence of an inflammasome associated to HS disease - Hypothesis It is widely accepted that hyperkeratinisation and follicular occlusion originate infection thereof causing skin inflammation. The investigators here hypothesized that host-derived danger signals led to the release of inflammatory mediators such as IL-1β by activating an inflammasome structure.

The inflammasome is a molecular platform controlling the expression and the activation of IL-1β via different sensors. The proinflammatory cytokine IL-1β could subsequently lead to the recruitment and orientation of lymphocytes towards a Th17 subtype creating a feedback loop maintaining excessive tissue inflammation in HS.

If such a complex inflammatory process is present in HS, blocking both the bacterial-induced (IL-1 β) and the sterile-associated (IL-17) inflammation would largely improve the therapeutic benefit for HS patients.

- Experimental approach

The investigators will seek to highlight the presence of inflammasome sensors and effectors in skin explants from HS compared to control skin. For this original physiopathological study, 10 lesional skins excised from HS patients or controls (plastic surgery) after they signed informed consent as required by the ethical review board (CPP accepted on the 23-01-2015) will be investigated. HS disease severity will be based on staging according to Hurley staging. Six mm skin punches will be harvested from control explants and from both in situ and peri-lesional sites of HS skin explants. Skin samples will be handled either straight forwardly (day 0) or after a period of tissue culture of 4 days with or w/out treatments.

All experiments will be conducted as follows:

* Ex vivo skin tissue samples will be inserted in a Transwell® filter and cultured over a period of 4 days with or w/out antibiotics (Rifampicin, Clindamycin).
* Both at day 0 and day 4:

  * one set of skin samples will be embedded to analyze the presence of inflammasome sensors and effectors by immunohistochemistry (IHC)
  * Another set will be homogenized for cytokines determination (ELISA) and cell stimulation (see below)
* Homogenized samples will be treated or not with anti-cytokine antibodies (Secukinumab vs isotype) for 4 hours before addition to keratinocytes cell line or monocyte/macrophage cell line. The influence of IL-17 and bacterial infection on inflammasome activation in these cell lines will be investigated as above described and associated with PCR technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe HS in the Dermatology department of Reims CHU, and eligible for surgery
* Patients accepting to participate to the study (signed consent)
* Patients affiliated to a certain social scheme
* Controls with plastic surgery but without HS, affiliated to a certain social scheme and accepting to participate

Exclusion Criteria:

* Patients <18yo

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2015-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
cytokine quantification (IL1-β) by ELISA | up to 4 days
cytokine quantification (IL-10) by ELISA | up to 4 days
cytokines quantification (IL-13) by ELISA | up to 4 days
cytokines quantification (IL-18) by ELISA | up to 4 days
cytokines quantification (CXCL10) by ELISA | up to 4 days
cytokines quantification (TNFα) by ELISA | up to 4 days
cytokines quantification (TGFβ) by ELISA | up to 4 days

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, France, Reims, France

REFERENCES:
- [Background] Sanchez J, Le Jan S, Muller C, Francois C, Renard Y, Durlach A, Bernard P, Reguiai Z, Antonicelli F. Matrix remodelling and MMP expression/activation are associated with hidradenitis suppurativa skin inflammation. Exp Dermatol. 2019 May;28(5):593-600. doi: 10.1111/exd.13919. PMID 30903721